CLINICAL TRIAL: NCT01910896
Title: A Prospective, Intra-individual Randomized, Observer-blind, Controlled Investigation to Investigate the Effectiveness and Safety of Overnight Intensive Patch (OIP) Over 12 to 24 Weeks in Post Dermatological Surgery Scars
Brief Title: Effectiveness and Safety Study of Overnight Intensive Patch in Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MRZ90011_0028_3
Record Dates: First submitted 2013-07-18; First posted 2013-07-30 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Post Dermatological Surgery Scars

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Overnight Intensive Patch (Experimental): Overnight intensive patch (OIP), on polyolefin foam basis containing acrylate, extractum cepae and allantoin is a class I, CE (Conformité Européenne) marked medical device. Subjects will have their two scars randomized for Overnight Intensive Patch application versus no treatment.
  Interventions: Device: Overnight Intensive Patch
- No treatment (No Intervention): Subjects serve as their own control. Eligible subjects have two comparable scars in same body regions, one scar will be treated with Overnight Intensive Patch, the second scar will not be treated.

INTERVENTIONS:
Device: Overnight Intensive Patch — Eligible subjects will have their two scars randomized for OIP application/no treatment. OIP for overnight application (at least 6 hours) for 12 to 24 weeks.
  Arms: Overnight Intensive Patch

SUMMARY:
To investigate the effectiveness of an Overnight Intensive Patch (OIP) on improvement of post dermatological surgery scars and its safety over 12 to 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject has two or more newly formed post dermatological surgery scars of 1-10 (inclusive) cm each, with comparable length, located on a comparable skin area (upon the discretion of the investigator, considering e.g. the skin thickness or body tension). Scars located at the upper back of the body will not be investigated due to a higher risk of wound dehiscence.
* The dermatological surgery takes place within the last 3 weeks prior to baseline visit and the baseline visit is on the day of post-surgery control with optional suture removal, the wound must be closed by then.

Exclusion Criteria:

* Subject with known history of keloids or hypertrophic scars.
* Subject with derma resurfacing procedures or non-invasive skin-tightening procedures including medium/ deep chemical peeling, dermabrasion treatments or laser therapy in the skin area intended to be treated for less than 8 weeks prior to screening/ baseline visit.
* Subject with any planned topical application containing active ingredients (e.g. self-tanning agents, however, hydration lotion is allowed provided the scars are left free) in the skin area intended to be treated.
* Subject anticipated spending excessive time in the sun (e.g. outdoor workers) or in the sun tanning bed during the investigation.
* Subject with any infection or wound in the area intended to be treated.
* Subject with known hypersensitivity to any ingredient of OIP (e.g. acrylic adhesive, extractum cepae or allantoin).
* Subject who is taking, or anticipated to take during the investigation, systemic corticosteroids or topical corticosteroids applied on the investigation skin area.
* Subject with eczema requiring treatment in the skin area intended to be treated.
* Subject with any ongoing severe or uncontrolled systemic disease (cardiac, respiratory, hepatic, renal or gastrointestinal), malignant tumor (except for basalioma), or known HIV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2013-10; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Absolute change from screening/baseline in the total score of observer evaluated POSAS [Patient and Observer Scar Assessment Scale] to week 12 | Baseline to week 12
  The POSA scale consists of two scales which need to be filled out by the observer and the subject, respectively. The scale will be rated for both scars of the same subject by observer and the subject independently in all planned visits.
  Observer Scar Assessment: The observer assesses the following items on a scale from 1 (normal skin) to 10 (worst imaginable skin): Vascularization, Pigmentation, Thickness, Relief, Pliability.
  Patient Scar Assessment: The subject answers the following questions on a scale from 1 (no, no complaints) to 10 (yes, worst imaginable): Is the scar painful?, Is the scar itching?; The subject answers the following questions on a scale from 1 (no, as normal skin) to 10 (yes, very different): Is the color of the scar different?, Is the scar more stiff?, Is the thickness of the scar different?, Is the scar irregular?

SECONDARY OUTCOMES:
Absolute change from screening/baseline in the total score of patient evaluated POSAS to week 12 | Baseline to week 12
Absolute change from screening/baseline in the total score of observer evaluated POSAS to week 24 | Baseline to week 24

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz Pharmaceuticals GmbH
Locations (9):
- Germany (9):
  - Merz Investigational Site # 0490341, Augsburg
  - Merz Investigational Site # 0490312, Berlin
  - Merz Investigational Site # 049307, Hamburg
  - Merz Investigational Site #0490345, Hamburg
  - Merz Investigational Site # 0490101, Mahlow
  - Merz Investigational Site #0490340, Mainz
  - Merz Investigational Site # 049112, München
  - Merz Investigational Site # 049331, Münster
  - Merz Investigational Site # 0490321, Schweinfurt